CLINICAL TRIAL: NCT04172233
Title: A Randomized, Double-blinded, and Placebo-controlled Phase I/II Clinical Study of AK101 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Clinical Study of AK101 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK101-101
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Plaque Psoriasis
Keywords: IL12/23

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Phase I: AK101 45 mg (Experimental): Biological: AK101 AK101 45 mg on Week 0 and 4 by subcutaneous injection
  Interventions: Biological: AK101
- Phase I: AK101 135 mg (Experimental): Biological: AK101 AK101 135 mg on Week 0 and 4 by subcutaneous injection
  Interventions: Biological: AK101
- Phase I: AK101 270 mg (Experimental): Biological: AK101 AK101 270 mg on Week 0 and 4 by subcutaneous injection
  Interventions: Biological: AK101
- Phase I: Placebo (Placebo Comparator): Biological: Placebo Placebo on Week 0 and 4 by subcutaneous injection
  Interventions: Biological: placebo
- Phase II: AK101 45 mg (Experimental): Biological: AK101 AK101 45 mg on Week 0, 4 and 16 by subcutaneous injection
  Interventions: Biological: AK101
- Phase II: AK101 90 mg (Experimental): Biological: AK101 AK101 90 mg on Week 0, 4 and 16 by subcutaneous injection
  Interventions: Biological: AK101
- Phase II: AK101 135 mg (Experimental): Biological: AK101 AK101 135 mg on Week 0, 4 and 16 by subcutaneous injection
  Interventions: Biological: AK101
- Phase II: Placebo to AK101 (Placebo Comparator): Drug: Placebo Placebo on Week 1 and 4 by subcutaneous injection, and then AK101 on Week 12 16 by subcutaneous injection
  Interventions: Biological: AK101; Biological: placebo

INTERVENTIONS:
Biological: AK101 — AK101 is an anti-IL-12/23p40 monoclonal antibody.
  Arms: Phase I: AK101 135 mg; Phase I: AK101 270 mg; Phase I: AK101 45 mg; Phase II: AK101 135 mg; Phase II: AK101 45 mg; Phase II: AK101 90 mg; Phase II: Placebo to AK101
Biological: placebo — matching placebo
  Arms: Phase I: Placebo; Phase II: Placebo to AK101

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and the preliminary efficacy of AK101，an anti-IL-12/23p40 monoclonal antibody, when administered subcutaneously in subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, placebo-controlled trial which consisted of a dose escalation phase (Phase I) and a dose expansion phase (Phase II)..

ELIGIBILITY:
Inclusion Criteria:

1. Have had Plaque Psoriasis diagnosed at least 6 months prior to screening.
2. Clinical diagnosis of stable plaque psoriasis with involvement of ≥ 10% body surface area. Psoriasis area and severity index(PASI) ≥12. Physicians Global Assessment score ≥3.
3. Patients who have received systemic therapy or phototherapy, or who have been allowed by the investigator to receive systemic therapy or phototherapy.
4. Women of childbearing potential should not be in pregnancy or lactation, men and women of childbearing potential must agree to use adequate birth control measures during study participation and for 6 months after the last dose of study treatment.
5. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.

Exclusion Criteria:

1. Had nonplaque forms of psoriasis (e.g., Guttate, erythrodermic, or pustular).
2. Had other active skin diseases or skin infections (e.g., bacterial, fungal or viral infection) that could affect psoriasis evaluation.
3. Had Imaging diagnosis of pulmonary infection or fibrosis during the 3 months prior to screening.
4. History or evidence of active or latent tuberculosis at screening.
5. Serious systemic infections or local infections during the 2 months prior to screening.
6. History of cancer, including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved).
7. Known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.
8. History of alcohol or drug abuse.
9. History or known presence of recurrent or chronic infection (e.g., hepatitis B, or C, human immunodeficiency virus [HIV], syphilis, TB).
10. Had received any DMARDs (e.g., anti-malaria drug, retinoids, interferon, lithium) during 2 weeks prior to screening.
11. Had received any physical therapy (e.g., PUVA, ultra-violet therapy, tanning beds) during 2 weeks prior to screening.
12. Had received any systemic psoriasis therapy (e.g., glucocorticoid, retinoids, ciclosporin, methotrexate, or tripterygium) during 4 weeks prior to screening.
13. Had Enrolled in any other trials during 3 months prior to screening or concurrently enrolled in any other trials.
14. Had received previous treatment with any anti-IL-12/IL-23, IL-12, IL-23, IL-17 therapy for the treatment of psoriasis or psoriatic arthritis.
15. Had received previous treatment with natalizumab or any other drugs that regulate B cells or T cells (rituximab, abatacept, alemtuzumab) during 12 months prior to screening.
16. Had received other biologic therapy (e.g., TNF inhibitor) during 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | From the time of signing informed consent till Week 16 for Phase I or Week 28 for Phase II

SECONDARY OUTCOMES:
Number of participants who achieved ≥ 75% reduction in Psoriasis Area and Severity Index (PASI75) | At Week 2, 4, 8, 12, 16, 20 (Phase II), 24 (Phase II) and 28 (Phase II)
Number of participants who achieved ≥ 90% reduction in PASI (PASI90) | At Week 2, 4, 8, 12, 16, 20 (Phase II), 24 (Phase II) and 28 (Phase II)
Change From Baseline in the Physician Global Assessment (PGA) | At Week 2, 4, 8, 12, 16, 20 (Phase II), 24 (Phase II) and 28 (Phase II)
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose till Week 16 for Phase I or Week 28 for Phase II
  The immunogenicity of AK101 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Area under the curve (AUC) of AK101 | From first dose till Week 16 for Phase I
  The endpoints for assessment of PK of AK101 include serum concentrations of AK101 at different timepoints after AK101 administration.
Minimum observed concentration (Cmin) of AK101 | From first dose till Week 16 for Phase I or Week 28 for Phase II
  The endpoints for assessment of PK of AK101 include serum concentrations of AK101 at different timepoints after AK101 administration.
Maximum observed concentration (Cmax) of AK101 | From first dose till Week 16 for Phase I or Week 28 for Phase II
  The endpoints for assessment of PK of AK101 include serum concentrations of AK101 at different timepoints after AK101 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Chen, MD, Principal Investigator — Peking Union Medical College Hospital; Hongzhong Jin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No